CLINICAL TRIAL: NCT04875936
Title: Rehabilitation of Reading Deficits in Subacute Stroke Using Functional Magnetic Resonance Imaging (fMRI) Neurofeedback and Motor Imagery
Brief Title: Neurofeedback Intervention for Reading Deficits in Subacute Stroke
Acronym: ReadingNFB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kessler Foundation (Other)
Responsible Party: Principal Investigator, Olga Boukrina, Research Scientist, Kessler Foundation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R-1147-21
Record Dates: First submitted 2021-04-29; First posted 2021-05-06 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Stroke; Dyslexia, Acquired
MeSH Terms: conditions — Stroke; Dyslexia, Acquired

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of 2 groups
Who Masked: Participant
Masking Description: Participants will be masked to the nature of real-time fMRI neurofeedback they will receive: contingent or non-contingent.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Motor Imagery and Contingent Neurofeedback (NFB) (Experimental): This group will receive real-time fMRI NFB on the bases of participant's own brain activity
  Interventions: Behavioral: Motor Imagery and Real-Time fMRI Neurofeedback
- Motor Imagery and Non-contingent Neurofeedback (NFB) (Sham Comparator): This group will receive group will receive fMRI NFB based on another participant's brain activity
  Interventions: Behavioral: Motor Imagery and Sham fMRI Neurofeedback

INTERVENTIONS:
Behavioral: Motor Imagery and Real-Time fMRI Neurofeedback — Survivors of left-hemisphere stroke (<10 weeks post-stroke) or healthy volunteers will use right-hand motor imagery coupled with fMRI neurofeedback to help them re-engage the left hemisphere by shifting brain activation leftward relative to the initial left-right asymmetry. Following group assignment, participants will perform a motor imagery task and complete 3 sessions of motor imagery and reading tasks in the MRI scanner over 3 weeks. During the MRI sessions they will receive real time neurofeedback about how well they are engaging the left side of their brain compared to the right side. They will also practice the same task for 30 min a day as homework using the most effective motor imagery strategy that worked for them in the MRI scanner.
  Arms: Motor Imagery and Contingent Neurofeedback (NFB)
Behavioral: Motor Imagery and Sham fMRI Neurofeedback — Survivors of left-hemisphere stroke (<10 weeks post-stroke) or healthy volunteers will practice right-hand motor imagery coupled with sham fMRI neurofeedback. As the experimental group, participants will perform a motor imagery task and complete 3 sessions of motor imagery and reading tasks in the MRI scanner over 3 weeks. However, during the MRI sessions they will receive sham neurofeedback on the basis of another participant's brain activity. Like the experimental group, they will also practice the same task for 30 min a day as homework.
  Arms: Motor Imagery and Non-contingent Neurofeedback (NFB)

SUMMARY:
The overall goal of this project is to advance a biologically-based approach to treatment of reading disorders after stroke, which will expand the limits of cognitive rehabilitation. Using a novel brain imaging technique, called real-time functional magnetic resonance imaging (fMRI) neurofeedback combined with right hand motor imagery, this project will re-instate brain activity in the left language-dominant hemisphere. Stroke patients will practice modulating their own brain activity using fMRI neurofeedback signal and will select the most effective mental strategies that help them maintain brain activation patterns associated with better reading recovery.

ELIGIBILITY:
Inclusion Criteria:

* First-ever left-hemisphere stroke < 3 months prior to study recruitment or healthy volunteer
* Age: 18 - 80 years old
* Fluent and literate in English prior to stroke
* Reading deficits, defined as >3 errors on the Paragraphs test (subtests VIII, IX) of the Reading Comprehension Battery for Aphasia-2nd ed. (RCBA-2) in keeping with the healthy control accuracy criterion of 86-100% correct.

Exclusion Criteria:

* Inability to consent or complete study tasks
* Inability to undergo MRI (e.g., pregnancy, non-MRI compatible implants, claustrophobia)
* A history of prior neurological disease (e.g., brain tumor, Alzheimer's disease)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2023-04-03 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Reading Aloud Accuracy | change from baseline at intervention week 1, 2, and 3
  Read aloud 136 words to produce an accuracy score in percent correct.
fMRI Brain Activity | change from baseline at intervention week 1, 2, and 3
  Whole-brain and region of interest activation and resting state functional connectivity

SECONDARY OUTCOMES:
Reading Comprehension Battery for Aphasia (RCBA-2) | change from baseline at 1 week follow up
  Letter, word, sentence, paragraph and text-level reading comprehension test designed for aphasia. Score range 0-100, higher scores correspond to better reading ability.
Western Aphasia Battery-Revised (WAB-R) Bedside | change from baseline at 1 week follow up
  A bedside assessment for language impairments in aphasia. Scores range from 0 to 80 for the Bedside Language Score and higher scores represent better language ability.
Boston Naming Test (BNT-short) | change from baseline at 1 week follow up
  A brief picture naming test designed to identify word finding difficulties. Score ranges from 0 to 15, with higher scores corresponding to better picture naming ability.
Palm Trees and Pyramids test | change from baseline at 1 week follow up
  Touch-screen computer tests of semantics, phonology, and orthography. The semantics task is to choose one of two examples at the bottom of the screen that matches the target at the top in meaning. The phonology task is to select a rhyme of the target in a similar fashion. These tests have a word and picture versions. The orthography task is to choose a letter string that more closely resembles a word. Each subtest accuracy ranges from 0 to 60 items, with higher scores representing better function.
Geriatric Depression Scale (GDS) | change from baseline at 1 week follow up
  A self-report assessment of depression to be used as covariate where appropriate. Scores range 0-30, with higher scores representing worse self-ratings of depression.
Neuro evaluation | baseline and 1 week follow up
  An in-house test of motor and cognitive function, administered by a qualified clinician. The test includes observational checklists, testing 9 qualitative parameters: mental status, cranial nerves, motor function, sensory function, reflexes, cerebellar function, gait and stance, behavior during testing and any other observations.

CONTACTS AND LOCATIONS:
Locations (1):
- Kessler Foundation, West Orange, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
Data generated in this project may be shared in accordance with the funding agency (NIH) and site organization (Kessler Foundation) policies, as well as the Notice of Privacy of Practices and Informed Consent documents signed by each participant in the study. In case data are shared, they will be de-identified, such that no link can be made to the individual participant. To prevent the possibility of deductive disclosure of participants through brain scans and the association with the rehabilitation hospital, data and associated documentation will be made available to users only under a data-sharing agreement.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Data may be shared after the acceptance for publication of the main findings of the study.
Access Criteria: Data may be shared upon request and following the establishment of a data sharing agreement, that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed.

REFERENCES:
- [Derived] Boukrina O, Yamin A, Yue GH, Kong Y, Koush Y. Feasibility of real-time fMRI neurofeedback for rehabilitation of reading deficits in aphasia. medRxiv [Preprint]. 2025 Jan 5:2025.01.03.25319980. doi: 10.1101/2025.01.03.25319980. PMID 39802782